CLINICAL TRIAL: NCT02293564
Title: An Open-label Safety Extension Study of Gevokizumab in Active Inflammatory, Erosive Osteoarthritis of the Hand
Brief Title: Open-label Safety Extension Study of Gevokizumab in Erosive Osteoarthritis of the Hand
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: XOMA (US) LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: X052161
Record Dates: First submitted 2014-11-11; First posted 2014-11-18 (Estimated); Last update posted 2015-02-19 (Estimated); Status verified 2015-02

CONDITIONS: Osteoarthritis
Keywords: Erosive Osteoarthritis; Osteoarthritis; Osteoarthritis of the Hand
MeSH Terms: conditions — Osteoarthritis | interventions — gevokizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- gevokizumab (Experimental)
  Interventions: Drug: gevokizumab

INTERVENTIONS:
Drug: gevokizumab — Solution for subcutaneous injection

SUMMARY:
The purpose of this study is to evaluate the long-term safety of gevokizumab in the treatment of active inflammatory, erosive osteoarthritis of the hand.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hand osteoarthritis
* Joint tenderness and/or redness
* At least one erosion by X-ray (as determined by the central reader)
* Contraceptive measures adequate to prevent pregnancy during the study

Exclusion Criteria:

* History of inflammatory disease other than hand erosive osteoarthritis (EOA) including: secondary post-traumatic osteoarthritis (OA); rheumatoid arthritis; spondylarthropathies; erosion of the ulnar styloid process; psoriatic arthritis; skin psoriasis; erosions of the wrist; fibromyalgia
* History of gout, pseudogout, or hemochromatosis
* History of allergic or anaphylactic reactions to monoclonal antibodies
* History of recurrent or chronic systemic infections
* Female subjects who are pregnant, planning to become pregnant, have recently delivered, or are breast-feeding

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2013-03; Primary Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Treatment-emergent adverse events | Up to two years
  Safety analyses will involve examination of the incidence, severity, and type of treatment-emergent adverse events reported.

CONTACTS AND LOCATIONS:
Locations (28):
- United States (28):
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Roseville, California
  - Sacramento, California
  - Santa Monica, California
  - Boulder, Colorado
  - Denver, Colorado
  - Miami, Florida
  - Pinellas Park, Florida
  - Tampa, Florida
  - Vero Beach, Florida
  - West Palm Beach, Florida
  - Indianapolis, Indiana
  - Wichita, Kansas
  - Hagerstown, Maryland
  - Wheaton, Maryland
  - Reno, Nevada
  - Albuerque, New Mexico
  - Raleigh, North Carolina
  - Portland, Oregon
  - Duncansville, Pennsylvania
  - Austin, Texas
  - Dallas, Texas
  - San Antonio, Texas
  - Waco, Texas
  - Charlottesville, Virginia
  - Norfolk, Virginia
  - Franklin, Wisconsin